CLINICAL TRIAL: NCT06101303
Title: The Mechanisms Underlying Endometriosis Pain
Brief Title: Endometriosis Pain
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Hadas Nahman-Averbuch, Asst Prof of Anesthesiology, Washington University School of Medicine
Other Study IDs: 202305023
Record Dates: First submitted 2023-10-02; First posted 2023-10-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Pain; Endometriosis
MeSH Terms: conditions — Pelvic Pain; Endometriosis | interventions — Blood Specimen Collection; Urination; Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometriosis lesions and/or peritoneal biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic pain: Patients with pelvic pain with and without endometriosis scheduled for an operative laparoscopic surgery for endometriosis diagnosis and/or treatment
  Interventions: Other: Psychophysical assessment; Behavioral: Psychophysical assessments of experimental pain; Diagnostic Test: Blood, urine and saliva samples; Procedure: Biopsy and surgery-related data.

INTERVENTIONS:
Other: Psychophysical assessment — Thermal stimuli: The Thermal Sensory Analyzer will be used to deliver heat and cold stimuli. All targeted stimulus temperatures will be less than 50°C, and participants will be free to remove their arm or leg at any time from the thermode. Noxious cold stimuli will also be delivered with a plastic water bath or an electronic electronic temperature-controlled water bath. Participants will be free to pull out of the water bath at any time.
  Pressure stimuli: Pressure stimuli will be applied by using a handheld algometer. These devices have a round probe that allows quantifying the amount of pressure that is being applied by real-time visual feedback to control and monitor applied pressure rates. Pressure will be applied to the lower leg, volar forearm, or trapezius.
  Mechanical stimuli: A set of standardised von Frey filaments (0.25, 0.5, 1, 2, 4, 8, 16, 32, 64, 128 and 256mN). The contact area of the hairs with the skin is of uniform size (<1 mm²) and texture.
Behavioral: Psychophysical assessments of experimental pain — Pain ratings- Pain intensity and pain unpleasantness ratings will be assessed
  Pain thresholds to heat, cold and/or pressure will be tested and participants will be instructed to press a button the first moment they feel pain.
  Temporal summation- participants will rate the pain evoked by a single pinprick stimulus and by a series of 10 identical pinprick stimuli.
  Conditioned pain modulation (CPM) efficiency - CPM testing includes the application of a "test" stimulus without conditioning (heat or pressure stimuli) and a subsequent application of the same test stimulus together with a conditioning stimulus (cold stimulus).
  Offset analgesia will be assessed using the three-temperature method (T1°C 5s, T1+1°C 5s, T1°C 20s). During the OA paradigm, real time pain intensity ratings will be obtained
  Cold pain tolerance will be assessed by having participants immerse their hand or foot in a cold water bath. Tolerance will be defined by the time of hand/foot withdrawal.
Diagnostic Test: Blood, urine and saliva samples — Blood (approximately 2 tablespoons), urine and saliva samples will be collected and sent to ZRT Laboratory, LabCorp, or internal Washington University lab for analyses of sex hormone levels (e.g., testosterone, estradiol, progesterone). Additional samples will be stored in a biobank for future processing.
Procedure: Biopsy and surgery-related data. — During the surgery, biopsies will be collected from the endometriosis lesions as well as from a healthy peritoneum. If there are no endometriosis lesions, biopsies will be taken of two common locations where endometriosis lesion grows (the infra-ovarian fossa). The lesions will be characterized based on their appearance and invasiveness of the lesions (i.e., powder-burn lesions, nonclassical red or white lesions, and superficially or deeply infiltrating (>5mm) lesions). In addition, surgery-related data such as the incision size, type of anesthesia, pain ratings after the surgery, analgesic medication after the surgery, and side effects will be documented. Blood, saliva, urine, and samples will be collected for hormonal analyses or stored in a Biobank for future analyses.

SUMMARY:
Aim 1. To determine the factors contributing to pain in patients with chronic pelvic pain with and without endometriosis Aim 2. To determine the changes following endometriosis lesion removal surgery in pain and sex hormone levels.

Aim 3. To identify factors predicting clinical pain reduction after lesion removal surgery.

Additional exploratory aims might compare subgroups of patients such as patients with vs. without endometriosis, with vs. without additional chronic pain syndromes, and with vs. without hormonal treatment. In addition, the role of lesion-specific immune signatures and psychological factors on pain will be explored.

Patients with pelvic pain potentially due to endometriosis will complete questionnaires including social, health, behavioral, and psychological questionnaires. Patients will also complete a 2.5 hours study visit of psychophysical assessments of thermal and pressure stimuli. In addition, blood, urine, and saliva samples will be collected for hormonal, immune, and genetic analyses. Additional samples might be collected and stored for future analyses. For some participants, these procedures will be completed several times, including before the surgery as well as 3 months, 6 months and 1 year after surgery. After the surgery, surveys assessing pain and other symptoms will be sent every week on the first month and then monthly for 1 year. In addition, during the surgery, biopsies will be collected and analyzed to determine hormonal, immune and genetic factors.

For adolescents, a parent/legal guardian will be asked to assist in completing some of the health-related surveys (i.e., physical developmental survey, health survey, migraine history survey).

DETAILED DESCRIPTION:
Pre-Study Period

Participants will be recruited via the pain and Ob/Gyn clinics and via EPIC. Potential participants might be identified via EPIC records using age, sex, diagnoses, notes, problem list, medications, date of scheduled surgery, name of physician performing the surgery, and phone number.

A research staff member will contact a potential participant and provide a description of the project. Potentially eligible participants will be invited to participate in the study, which will be conducted at Washington University School of Medicine. Participants will also be provided with a written summary or the consent of the study. The consent will be signed electronically, using Docusign e-consent process or remotely during a phone call or a video call (WUSTL Zoom) with a study staff or in person.

Study Design

After confirming the inclusion criteria and signing the consent form, patients with pelvic pain potentially due to endometriosis will complete a 2.5 hours study visit of psychophysical assessments of thermal and pressure stimuli. Patients will also complete various questionnaires including demographic, social, health, behavioral, and psychological questionnaires. . For adolescents, a parent/legal guardian will be asked to assist in completing some of the health-related surveys (i.e., physical developmental survey, health survey, migraine history survey). Obstetric, gynecologic, fertility, and surgical history will be abstracted from the medical record and/or via health history interview. These procedures will be completed before the surgery.

During the surgery, the endometriosis lesions will be excised as part of routine care. At least one lesion will be sent to pathology and one lesion for the study team. In the absence of lesions, peritoneally biopsies of bilateral infra-ovarian fossa will be collected per routine practice. One will be sent to pathology, and one for the study team. Vials of health abdominal peritoneum, and endometrial biopsy (if uterus present) will be collected for study purpose.

Before or on the day of the surgery, blood, urine, and/or saliva samples will be collected for hormonal, immune and genetic testing. Additional samples will be stored in a biobank for future hormonal, immune and/or genetic analyses.

In addition, after the surgery, participants will be asked to complete surveys assessing pain and other symptoms which will be sent every week for the first month and then monthly for 1 year.

After the surgery, participants will have the option to return for additional study visits that will include the same psychophysical procedures and collection of blood (about 20 ml), urine, and/or saliva samples (3 months, 6 months and 1 year after surgery).

During the study period, new about pelvic pain, new/changes in diagnosis, treatment changes (medication titration, physical therapy, mental health, and alternative therapies), surgery related data, additional pain-related diagnoses, and additional markers (i.e., vitamin D, hormone levels) will also be collected via EPIC and/or health history interview.

All study procedures are optional and participants can stop or not complete tests if they want.

Participants need to meet all the inclusion criteria to be included in the study. After consenting and the first study visit, changes in health will not automatically lead to excluding participants from the study. Before the follow-up visits, the investigators will ask the participants about changes in their health (from the last visit). Based on the responses, continuation/withdrawal from the study and/or omission of study activities will be determined at the discretion of the PI and/or study staff.

ELIGIBILITY:
Inclusion criteria:

* Patients with pelvic pain with and without endometriosis scheduled for an operative laparoscopic surgery for endometriosis diagnosis and/or treatment
* Age 12-45
* Females

Exclusion criteria:

* Pregnancy
* Planned hysterectomy or oophorectomy
* Co-occurring vaginismus and/or vulvodynia
* For patients aged 12-17 not having a parent/legal guardian willing to sign the consent and answer surveys about their child's health

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Female patients with pelvic pain scheduled for an operative laparoscopic surgery for endometriosis diagnosis and/or treatment
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain ratings of clinical pain | Baseline and follow up (3 months, 6 months and 1 year after surgery)
  Rating the pain intensity level using a numerical pain scale (0-100) or visual analog scale
Estrogen levels | Baseline
  systemic estrogen level and local estrogen level from the lesion
Estrogen receptor expression in the lesion | Baseline
  analyzing the levels of estrogen receptor expression in the endometriosis lesion
Conditioned pain modulation (CPM) response | Baseline and follow up (3 months, 6 months and 1 year after surgery)
  The CPM paradigm assesses endogenous inhibitory pain modulation efficiency. CPM testing includes the application of a "test" stimulus without conditioning (control run, pressure pain thresholds) and a subsequent application of the same test stimulus together with a conditioning stimulus (conditioning run, a 60 second of foot immersion in cold water). The CPM response is the difference in the pressure pain thresholds between the control and the conditioning runs.

SECONDARY OUTCOMES:
Pressure pain thresholds (PPT) | Baseline and follow up (3 months, 6 months and 1 year after surgery)
  Pressure will be increased continually and participants will be instructed to press a button the first moment they feel pain from the pressure stimulus. The first threshold measurement will be used as a familiarization. The average threshold is calculated from three measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Nahman-Averbuch, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No